CLINICAL TRIAL: NCT00590538
Title: A Pilot Trial of Phenylbutyrate/Genistein Duotherapy in Delta F508-Heterozygous Cystic Fibrosis Patients
Brief Title: Phenylbutyrate/Genistein Duotherapy in Delta F508-Heterozygotes (for Cystic Fibrosis)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 12/15/2008 Voluntarily placed on inactive status-requested by the PI
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Ronald Rubenstein, M.D., PhD., The Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2002-10-3023; RUBENS01A0 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2007-12-27; First posted 2008-01-10 (Estimated); Results first posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — 4-phenylbutyric acid; Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenylbutyrate (Active Comparator): The standard oral adult dose is 20 g/day for 4 days.
  Every participant will receive Genistein during the NPD.
  Interventions: Drug: Sodium 4-Phenylbutyrate; Drug: Genistein (Unconjugated Isoflavones 100)
- Placebo (Placebo Comparator): The placebo is given to match the active comparator for 4 days. Every participant will receive Genistein.
  Interventions: Drug: Genistein (Unconjugated Isoflavones 100); Drug: Placebo

INTERVENTIONS:
Drug: Sodium 4-Phenylbutyrate — The standard oral adult dose is 20 g/day (tablets) for 4 days.
  Other Names: 4PBA
  Arms: Phenylbutyrate
Drug: Genistein (Unconjugated Isoflavones 100) — Every participant will be administered a perfusion of 50 MicroM of Genistein (Unconjugated Isoflavones 100) during the modified NPD procedure.
  Other Names: PTI G-4660, 87% Genistein
Drug: Placebo — The placebo is given to match the active comparator for four days.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test a new combination of medicines, Phenylbutyrate and Genistein, to determine if they could be used to treat cystic fibrosis (CF). The most common genetic mutation found in patients with CF is called Delta F508. Due to this mutation, there is a lack of salt (chloride) movement in your nose, sinuses, lungs, intestines, pancreas and sweat glands. This lack of movement causes the clinical manifestations of the disease.

Although Phenylbutyrate has been extensively used to treat patients with rare metabolic diseases, Phenylbutyrate is an investigational drug for the purpose of this study. Genistein is a naturally occurring substance that is found in food products such as soy and tofu, but is also an investigational drug for this study. When used together, both drugs may be able to restore normal chloride and salt (water) movements in body organs and glands in people with CF.

We will be studying salt and water movement in the nose by a technique called nasal transepithelial potential difference (NPD).

DETAILED DESCRIPTION:
This protocol is investigating novel pharmaceutical agents (Phenylbutyrate and Genistein), which are aimed at improving the physiologic function of mutant Cystic Fibrosis Transmembrane conductance Regulator (CFTR). CFTR is absent or dysfunctional in cystic fibrosis. Nasal epithelial CFTR function will be assessed by the NPD procedure.

We will test the hypotheses that:

1. Phenylbutyrate given orally for 4 days will be safe in adult Delta F508- heterozygous subjects with CF and will result in small improvements in nasal epithelial CFTR function.
2. Topical administration of Genistein to the nasal epithelia of Phenylbutyrate treated Delta F508-heterozygous CF subjects will be safe and lead to augmentation of the improved nasal epithelial CFTR function observed during Phenylbutyrate treatment, but not during placebo treatment.

Study Flow If eligibility is confirmed at the screening visit, there will be an additional 3 outpatient visits over a 1-2 week period, lasting 2-4 hours each.

Visit 1, all study related safety evaluations will be completed. There will also be a Nasal Potential Difference (NPD) measurement performed. To measure nasal potentials, or voltages, a small butterfly needle will be placed in the skin of the forearm and connected by a thin plastic tube to a monitoring device. A very small soft plastic catheter or tube will be placed against the inner surface of the nose. This catheter will pump a very small amount of saltwater onto the nose and it will connect to the monitoring machine. This machine senses very small electrical voltages that are generated by the body. It does not and cannot send electricity or shocks to the subject. A measurement is made and then the fluid pumped into the nose is changed to one containing a drug called amiloride. Amiloride changes the makeup of salt transported in the nose and reduces the electrical voltage. Then the fluid is changed to saltwater that does not contain chloride. The fluid is then changed to one that has the drug isoproterenol. Isoproterenol causes the cells in subjects without CF to move chloride. The doses of amiloride and isoproterenol used in this study are much lower than those typically used in patients for other reasons. Finally, the fluid will be changed to one containing the experimental drug Genistein.

Subject will then be randomized and given a 4-day supply of the study drug.

Visit 2, subject will have safety evaluations and NPD performed in the same manner as previous visit. No more study drug after this visit.

Visit 3, subject will have safety evaluations and NPD performed without the perfusion of Genistein.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate with pertinent staff, able to understand and willing to comply with the requirements of the trial, and able and willing to give informed consent.
2. Willing to practice a reliable and study-accepted method of contraception during the study.
3. Diagnosis of cystic fibrosis consisting of both:

   1. clinical manifestations of cystic fibrosis and
   2. either cystic fibrosis genotype heterozygous for Delta F508 with a second identified CFTR mutation, or cystic fibrosis genotype with one Delta F508 allele and one unidentified allele and sweat sodium or chloride > 60 mEq/L
4. Oxyhemoglobin saturation greater than or equal to 92% while breathing room air

Exclusion Criteria:

1. Underlying diseases likely to limit life span and/or increase risk of complications:

   1. Cancer requiring treatment in the past 5 years, with the exception of cancers that have been cured, or in the opinion of the investigator, carry a good prognosis such as non-melanoma skin cancer, papillary thyroid carcinoma, and cervical cancer in situ.
   2. GI disease

   i. Inflammatory bowel disease requiring treatment in the past year ii. elevations in ALT or AST levels to greater than 3 times the upper limit of normal
2. Conditions or behaviors likely to affect the conduct of the study

   1. Current or anticipated participation in another intervention research project
   2. Recent (with 2 months) sinus surgery or nasal polypectomy
   3. Currently pregnant or less than 3 months post-partum
   4. Currently nursing or within 6 weeks of having completed nursing
   5. Unwilling to undergo pregnancy testing or to report possible or confirmed pregnancy promptly during the course of the study
   6. Unwilling to use a reliable contraceptive method for two months after the completion of the study.
   7. Major psychiatric disorder, which, in the opinion of the investigators, would impede conduct of the study, e.g., alcoholism
   8. Other condition, which, in the opinion of the investigators, would impede conduct of the study.
3. Glucocorticoids other than topical, ophthalmic, and inhaled preparations.
4. Conditions that would place the patient at an increased risk for complications:

   1. Pneumothorax within the last 12 months
   2. Uncontrolled diabetes
   3. Asthma or allergic bronchopulmonary aspergillosis requiring systemic glucocorticoid therapy within the last two months
   4. Sputum culture growing a pathogen that does not have in vitro sensitivity to at least two types of antibiotics which could be administered to the patient
   5. History of major hemoptysis: (Greater than 240 mL of blood within a 24-hour period within the last 12 months).
5. Medication use or conditions not specifically mentioned above, including severe or end stage CF lung disease, that may serve as criteria for exclusion at the discretion of the investigators.
6. History of significant cardiovascular disease, such as myocardial infarction, congestive heart failure, unstable arrhythmia, or uncontrolled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2003-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Rubenstein, M.D., PhD., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was terminated by the PI before completing enrollment
Groups:
- Phenylbutyrate or Placebo: Subjects will be randomized to receive either the Phenylbutyrate or placebo tablets for 4 days.
  PLEASE NOTE: AT THE TIME OF TERMINATION BY PI, THE STUDY WAS NOT UNBLINDED SO IT IS NOT KNOWN WHICH PARTICIPANTS WERE ASSIGNED TO WHICH GROUP.
  Every participant will receive Genistein during the Nasal Potential Difference (NPD).
Period: Overall Study
Arm/Group | Phenylbutyrate or Placebo
Started | 9 (STUDY NOT UNBLINDED AT TIME OF TERMINATION; THEREFORE NUMBER ASSIGNED TO EACH GROUP IS NOT KNOWN.)
Completed | 7
Not Completed | 2
Not completed — Study terminated before completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Voltage (mVolt) in Nasal Epithelium
Description: The basis of analysis for the primary outcome measure will be the comparison of data from both the standard CF Nasal Potential Difference (NPD) Protocol compared to a modified NPD protocol including the perfusion of Genistein.
  The NPD response will be compared from baseline to after study drug. NPD responses will then be compared between the Phenylbutrate group and the placebo group.
Time Frame: Baseline and 2 weeks
Population: No analysis was completed on data collected; AND study was never unblinded therefore details not available.
Measure: Number; unit: mVolts
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in FEV1 (Forced Expiratory Volume in 1 Second) in Spirometry.
Description: Outcome measure will be obtained from standard Pulmonary Function testing.
Time Frame: baseline and 2 weeks
Population: No analysis was completed on data collected.
Measure: Number; unit: Liters
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in FVC (Forced Vital Capacity)in Spirometry.
Description: Outcome measure will be obtained from standard Pulmonary Function testing.
Time Frame: baseline and 2 weeks
Population: No analysis was completed on data collected.
Measure: Number; unit: Liters
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse Events will be assessed and outcome measure obtained by completion of Interval history, physical and mental status examinations of every participant.
Time Frame: up to 2 weeks
Measure: Number; unit: participants
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Abnormal Laboratory Safety Tests
Description: Outcome measure will be obtained by completion of routine metabolic and hematological laboratory parameters for every participant. Metabolic testing willl include a CMP (comprehensive metabolic panel, ALT (alanine aminotransferase test), GGT (gamma-glutamyl transpeptidase), and Uric Acid; Hematological testing will include a complete blood count (CBC), and partial thromboplastin (PT/PTT).
Time Frame: up to 2 weeks
Population: No analysis was completed on data collected; More clinically efficacious compounds have been identified which suggested that completion of this study might not be as critical as when initially proposed; therefore, the study was terminated by PI.
Measure: Number; unit: participants
Arm/Group | Phenylbutyrate or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Phenylbutyrate or Placebo
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
No analysis was completed on data collected; More clinically efficacious compounds have been identified which suggested that completion of this study might not be as critical as when initially proposed; therefore, the study was terminated by PI.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No